CLINICAL TRIAL: NCT02437578
Title: Development of Clinical Tests to Predict the Success of Assisted Reproductive Techniques in a Fertility Clinic
Brief Title: Clinical Tests to Predict the Success of Assisted Reproductive Techniques
Status: Completed | Type: Observational
Sponsor: Martin Blomberg Jensen (Other)
Collaborators: Dansk Fertilitetsklinik (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: CBG study3
Record Dates: First submitted 2015-04-16; First posted 2015-05-07 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Infertility
Keywords: vitamin d; fertility; markers; endocrine disruption; reproduction
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Not number of subject but number of cycles/treatments Serum Seminal plasma follicular fluid DNA granulosa cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Infertile couples: Infertile couples referred to Dansk fertilitetsklinik (Danish Fertility clinic) for IUI, IVF and ICSI treatment

SUMMARY:
Today, it is evident that vitamin D has more widespread effects than the classical actions related to bone mineralization and calcium homeostasis. Vitamin D deficiency results in impaired reproductive performance in various species of animals, and recently the investigators have shown that the Vitamin D receptor (VDR), activating (CYP2R1, CYP27A1, CYP27B1) and inactivating (CYP24A1) enzymes are expressed in the human testis, epididymis, seminal vesicle, prostate and spermatozoa. Functional studies showed that activated vitamin D increases intracellular calcium and sperm motility in mature spermatozoa, and hence may be important not only for spermatogenesis but also for sperm function. Any test that might assist in guiding the treatment of the infertile couple would be beneficial both for most infertile couples and the society in general. The fact that vitamin D may play a role for human semen quality are now being tested clinically. If vitamin D supplementation proves efficient this opens for the first time for a causal, safe and cheap treatment of at least some cases of "idiopathic" impaired semen quality. This may also have consequences in the in vitro setting as activated vitamin D may be used to select high quality sperm during assisted reproductive techniques. The presence of the vitamin D receptor and vitamin D metabolizing enzyme CYP24A1 in particular is able to discriminate spermatozoa from normal and infertile men. CYP24A1 is expressed at the annulus of normal sperm, but it is virtually absent from spermatozoa from infertile men. This indicates that CYP24A1 expression may assist in predicting the chance of success by using insemination (IUI), IVF or ICSI. CYP24A1 expression is induced by activated vitamin D, which indicates that other VDR activated genes also may serve as positive predictive markers of fertility. In addition, vitamin D metabolites and other factors in the female reproductive tract will be measured to determine if they alone or in combination with other markers can determine whether the best solution for the infertile couple would be to do IUI, IVF, or ICSI. The suggested clinical trial may therefore be able to evaluate several secondary endpoints in addition to CYP24A1 in our search for predictive markers for fertilization. For instance several biomarkers in serum, seminal plasma or follicular fluid in conjunction with genetic polymorphisms in several genes important for reproductive function.

DETAILED DESCRIPTION:
Background Today, it is evident that vitamin D has more widespread effects than the classical actions related to bone mineralization and calcium homeostasis. Vitamin D deficiency results in impaired reproductive performance in various species of animals, and recently the investigators have shown that the vitamin D receptor (VDR), activating (CYP2R1, CYP27A1, CYP27B1) and inactivating (CYP24A1) enzymes are expressed in the human testis, epididymis, seminal vesicle, prostate and spermatozoa. Functional studies showed that activated vitamin D increases intracellular calcium and sperm motility in mature spermatozoa, and hence may be important not only for spermatogenesis but also for sperm function. A cross sectional study of 300 young healthy Danish men showed that men with lower levels of serum 25-hydroxyvitamin D have significantly lower number of normally developed and motile spermatozoa. Hitherto, most cases of male infertility have been classified as "idiopathic", and infertile couples have been referred to symptomatic treatment at infertility clinics. These fertility treatments are often physically demanding for the female partner as well as expensive for the health care system. Any test that might assist in guiding the treatment of the infertile couple would be beneficial both for the infertile couples and the society in general. Our findings that vitamin D may play a role for human semen quality are now being tested clinically. If vitamin D supplementation proves efficient this opens for the first time for a causal, safe and cheap treatment of at least some cases of "idiopathic" impaired semen quality. This may have consequences as vitamin D may be used to select high quality sperm during assisted reproductive techniques. The presence of the vitamin D receptor and vitamin D metabolizing enzymes in a particular CYP24A1 is able to discriminate sperm from normal and infertile men. CYP24A1 is expressed at the annulus of normal sperm but is virtually absent from spermatozoa from infertile men. This indicates that CYP24A1 may be used as a marker to discriminate between good and unhealthy sperm and may therefore serve as a predictive clinical marker for fertility. This indicates that CYP24A1 expression also may assist in predicting the chance of success by using insemination (IUI), IVF or ICSI. CYP24A1 expression is induced by activated vitamin D through the VDR, which indicates that other VDR activated genes also may serve as positive predictive markers of fertility.

In addition to the simple use of VDR, CYP24A1 and other vitamin D regulated genes in human sperm as clinical markers, it is also important to determine the function of vitamin D in reproduction. In order to understand this, it is important to determine the concentration of vitamin D metabolites in the male and female reproductive tract. For instance if vitamin D metabolites are undetectable in the male reproductive tract but measurable in the female reproductive tract then it may be important for signaling to the capacitated (activated) spermatozoa. The different vitamin D metabolites and other factors in the female reproductive tract will be measured to determine if they alone or in combinaton with other markers may be good predictors of the success following IUI, IVF, or ICSI treatment. The suggested clinical trial may therefore be able to evaluate several secondary endpoints in addition to CYP24A1 in our search for predictive markers for fertilization. For instance several biomarkers in serum, seminal plasma or follicular fluid in conjunction with known polymorphisms in several genes important for reproductive function. For instance genetic variation in FSH signaling. Single nucleotide polymorphisms (SNPs) related to genes encoding the FSHβ subunit (FSHB) and the FSH receptor (FSHR) affect FSH production (FSHB c.-211 G>T) and sensitivity/expression of its receptor in vitro (FSHR c.2039A>G & FSHR c.-29G>A). FSHR c.2039A>G, but not FSHR c.-29G>A, is associated with increased FSH levels in adult women, while there are conflicting results on FSHB c.-211 G>T (7;8). May these polymorphisms and other specific polymorphisms affect male and female fertility potential, semen quality and reproductive hormones.

SETTING, SCIENTIFIC PLAN AND RECRUITMENT Participants will be included among infertile couples referred for IUI, IVF or ICSI at Dansk fertilitetsklinik. The design is a prospective, blinded, single center cohort study. The investigation of all samples will be blinded since investigators have no information about the clinical data, treatment failure/succes. all participants will be followed until 9 months after their treatment to evaluate live birth rate, abortions etc.

PARTICIPANTS All referred infertile couples will be invited to participate, however both partners should be > 18 years and the women < 43 years old. women using donorinsemination will also be included. Anticipated 800-1000 IUI and 400 IVF/ICSI will be conducted at the clinic in the study period. The investigators assume that up to 600 IUI and 200 IVF/ICSI wish to participate. Thus, 800 treatments is the target for inclusion in the study. The investigators expect a small retraction rate (< 20) because of high motivation and no adverse effects.

ANALYSIS Reproductive hormones, genetic analyses, endocrine disrupters and growth factors will be analyzed at dept. of GR,Rigshospitalet and calcium regulators including vitamin D metabolites at Holbæk hospital.

SAMPLE SIZE CALCULATION AND STATISTICS The power estimate is based on the published data on CYP24A1 as a positive marker of semen quality. The association between clinical pregnancy and CYP24A1 is estimated to be comparable with the association with sperm motility. This imply that N=600 IUI will be enough to evaluate the effect of CYP24A1 as a marker of pregnancy and live birth rate because the investigators estimate that at least 12% will have a positive pregnancy test. When the inital collection of raw semen/percoll separated sperm and data have been completed an additional amount of clinical observations will be obtained after 9 months on live birth rate, abortions etc. Secondary analyses on the putative association between clinical endpoints and the expression of VDR and other Vitamin D regulated genesin sperm will be investigated on a randomly selected subset of samples N=300. All the listed genetic analyses will be conducted on all men and all the women with DNA. Follicular fluid will be collected during IVF or ICSI when there is no contamination with blood. Analyses of different markers in the follicular fluid and cells will be associated with oocyte quality, pregnancy and live birth rate.

ETHICS AND SIDE EFFECTS All the patients will have finished their inital visit and investigations, before they are invited to participate in the study. The loss of spermatozoa for each man as a result of making the cytospin will not influence the successrate of IUI, IVF or ICSI because the investigators will take less than 2.5% of the sperm pool.

PUBLICATION OF RESULTS All results, positive or negative will be submitted to peer reviewed scientific journals. Data will successively be obtained and transferred to a statistical database.

Predefined subgroup analyses Female age, sperm concentration, TTP, BMI, expression of CYP24A1/VDR in sperm, raw semen verus percoll separated, serum vitamin D levels and the listed genetic polymorphisms under secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* part of an infertile couple
* > 18 years of age

Exclusion Criteria:

* women >43 years of age
* men with sperm concentration < 0.1 million/ml

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All infertile couples referred to Dansk Fertilitetsklinik will be invited to participate. Anticipated 800-1000 IUI and 400 IVF/ICSI will be conducted during the planned study period. The investigators assume that up to 600 IUI and 200 IVF/ICSI wish to participate. Thus 600-800 treatments is the estimated target for inclusion in this study. The investigators expect a small retraction rate (< 20) because of high motivation and no adverse effects.
Sampling Method: Probability Sample
Enrollment: 542 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-10 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
CYP24A1 expression in sperm as a positive predictive marker of the number of pregnancies and live births following IUI | 9 months after semen analysis
  CYP24A1 expression is evaluated in the semen sample used for IUI

SECONDARY OUTCOMES:
CYP24A1 expression in sperm as a positive predictive marker of the number of pregnancies and live births following IVF/ICSI | 9 months after semen analysis
  CYP24A1 expression is evaluated in the semen sample used for IVF/ICSI
CYP24A1 expression in sperm as a positive predictive marker of the fertilization rate and blastocyst/4cell quality following IVF/ICSI | within 28-35 days from CYP24A1 expression
  CYP24A1 expression is evaluated in the semen sample used for IVF/ICSI
CYP24A1 expression as a better predictor of success by using IUI, IVF and ICSI than semen analysis | One month after semen analysis
  CYP24A1 expression is evaluated in the semen sample used for IUI/IVF/ICSI
VDR expression in sperm as a positive predictive marker of the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
  VDR expression is evaluated in the semen sample used for IUI/IVF/ICSI
VDR expression in sperm as a positive predictive marker of the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
  VDR expression is evaluated in the semen sample used for IUI/IVF/ICSI N300
RANKL expression in sperm as a positive predictive marker of the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
  VDR expression is evaluated in the semen sample used for IUI/IVF/ICSI N300
Expression of a vitamin D regulated gene in sperm as a positive predictive marker of the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
  Expression of a vitamin D regulated gene will be evaluated in the semen sample used for IUI/IVF/ICSI N300
Combined expression of CYP24A1, VDR and RANKL in sperm as a positive predictive marker of the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
  Expression the selected genes will be evaluated in the semen sample used for IUI/IVF/ICSI N300
CYP24A1, VDR and RANKL as markers for good quality sperm and progressive motile sperm. | day 1
  CYP24A1 and semen quality
Serum vitamin D determine expression of CYP24A1, VDR and RANKL in sperm | day 1
  associations between local expression and serum vitamin D
Serum levels of vitamin D metabolites as markers of good semen quality and higher chance of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
High serum level of OPG as markers of good semen quality and more pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
Serum level of RANKL as markers of low semen quality and low chance of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
Serum level of FGF23 and or Klotho as positive predictors of semen quality and the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
Serum level of LHCGRas a negative predictor of semen quality and the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
Serum level of total, undercarboxylated or matrix osteocalcin as markers of semen quality and the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
Serum levels of vitamin D regulated genes as markers of semen quality and the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
Serum levels of calcium and phosphate and semen quality and the number of pregnancies and/or live births following IUI, IVF, ICSI | 9 months after semen analysis
vitamin D metabolites in follicular fluid as a positive predictive marker of oocyte quality, fertilisationrate, implantation, pregnancy and/or live births following IVF/ICSInumber of pregnancies and/or live births following IUI, IVF, ICSI | 1 and 9 months after semen analysis
Concentration of calcium and phosphate in follicular fluid as a positive predictive marker of oocyte quality, fertilisationrate, implantation, pregnancy and/or live births following IVF/ICSI | 1 and 9 months after semen analysis
Concentration of 1,25 dihydroxyvitamin D in follicular fluid as a positive predictive marker of the probability of the CYP24A1 positive sperm to fertilize the oocyte and/or live births following IVF/ICSI | within 1 month after semen analysis and 9 months after semen analysis
Concentration of reproductive factors in follicular fluid as a positive predictive marker of with oocyte quality, fertilisationrate, implantation, pregnancy and/or live births following IVF/ICSI | 1 and 9 months after semen analysis
  Klotho, LHCGR TRAP5, calcium, phosphat,
Concentration of selected bone factors in follicular fluid as a positive predictive marker of with oocyte quality, fertilisationrate, implantation, pregnancy and/or live births following IVF/ICSI | 1 and 9 months after semen analysis
  RANKL, OPG, RANK, FGF23, Osteocalcin, MGP, DKK, calcitonin, PTHrP, SOST, Capthepsin K
Polymorphisms in the selected vitamin D regulated genes and semen quality, male reproductive hormone levels or pregnancy and/or live births following IUI/IVF/ICSI | 1 and 9 months after semen analysis
  VDR, CYP24A1, CYP2R1, RANKL, TRPV6, TRPV5, CatSper, CaSR, Osteocalcin, MGP, or other vitamin D regulated genes
Polymorphisms in the selected bone-gonadal genes and semen quality, male reproductive hormone levels or pregnancy and/or live births following IUI/IVF/ICSI | 1 and 9 months after semen analysis
  RANK, OPG, LHCGR, FGF23, Klotho, GPRC6a, PHEX, MEPE, DMP1,DKK1,PTHR, calcitonin, PTHrP, SOST, Capthepsin K, FSH, FSHR, SLC34A1-3, PIT1-2
Polymorphisms in selected gonadal genes and oocyte quality, AMH levels, female reproductive hormone levels or pregnancy and/or live births following IUI/IVF/ICSI | 1 and 9 months after semen analysis
  VDR, CYP24A1, CYP2R1, LHCGR, TRPV6, TRPV5, CatSper, GPRC6a, LHCGR, PHEX, MEPE, DMP1,DKK1,PTHR, PTHrP, FSH, FSHR, SLC34A1-3, PIT1-2 or other vitamin D regulated genes
Polymorphisms in selected bone genes and oocyte quality, AMH levels, female reproductive hormone levels or pregnancy and/or live births following IUI/IVF/ICSI | 1 and 9 months after semen analysis
  RANKL, OPG, FGF23, Klotho, CaSR, RANK, Osteocalcin, MGP, calcitonin, PTHrP, SOST, Capthepsin K
FSH signalling polymorhisms and reproductive function in women and men | 1 and 9 months after semen analysis
  Single nucleotide polymorphisms (SNPs) related to genes encoding the FSHβ subunit (FSHB) and the FSH receptor (FSHR) affect FSH production (FSHB c.-211 G>T) and sensitivity/expression of its receptor in vitro (FSHR c.2039A>G & FSHR c.-29G>A) FSHR c.2039A>G, but not FSHR c.-29G>A, is associated with increased FSH levels in adult women, while there are conflicting results on FSHB c.-211 G>T.
Endocrine disrupting chemicals in serum, follicular fluid, seminal fluid as predictive markers of semen quality, pregnancies and live birth rate following IUI, IVF, ICSI | 1 and 9 months after semen analysis
  * p,p'-DDE
  * Nonylphenol
  * Triclosan
  * Homosalate
  * Benzyl butyl phthalate
  * OD-PABA
  * Di-iso-butyl phthalate
  * Dibutyl phthalate
  * 4-Methylbenzophenone
  * Octyl methoxycinnamate
  * Benzophenone-3
  * Perfluorooctanoic acid
LHCGR i follicular fluid and serum as predictors of serum levels of sex hormones and gonadotropins | at the time for oocyte retrieval
  LHCGR measured in serum and follicular fluid from women undergoing IVF and ICSI
LHCGR as predictors of a responsiveness (number of follicles, collected oocytes, fertilisation, number of 2 and 4 cell embryos, and implantation) to hormonal treatment given during ART (hCG, Lh, FSH) | LHCGR at the time for oocyte retrieval and outcomes determined i the following week
  LHCGR measured in serum and follicular fluid from women undergoing IVF and ICSI.
LHCGR i follicular fluid and serum as predictors of oocyte quality, abortion rate and live birth rate | at the time for oocyte retrieval and up to nine months later
  LHCGR measured in serum and follicular fluid from women undergoing IVF and ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Jensen, MD, DMSc, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Dansk Fertilitetsklinik, Frederiksberg, Denmark

REFERENCES:
- [Derived] Wulff SM, Jorsal MJ, Kooij I, Krog H, Bentin-Ley U, Blomberg Jensen M, Yahyavi SK. Phosphate concentrations in follicular fluid during assisted reproductive treatment: relevance for ovarian function and fertility outcomes. Reprod Biol Endocrinol. 2025 May 14;23(1):69. doi: 10.1186/s12958-025-01408-w. PMID 40369590